CLINICAL TRIAL: NCT07264959
Title: An Observational Study in Patients With Indolent Systemic Mastocytosis
Brief Title: An Observational Study in Participants With Indolent Systemic Mastocytosis (ISM)
Status: Not yet recruiting | Type: Observational
Sponsor: Blueprint Medicines Corporation (Industry)
Responsible Party: Sponsor
Other Study IDs: BLU-285-2406
Record Dates: First submitted 2025-11-24; First posted 2025-12-04 (Actual); Last update posted 2025-12-04 (Actual); Status verified 2025-11

CONDITIONS: Indolent Systemic Mastocytosis
Keywords: ISM; Avapritinib; BLU-285; Selective KIT mutation-targeted tyrosine kinase inhibitor; Tyrosine kinase inhibitor; Mastocytosis; Neoplastic mast cells
MeSH Terms: conditions — Mastocytosis, Systemic; Mastocytosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — With the participant's informed consent and as approved by local IRBs/IECs, de-identified biological samples may be stored at a biosample repository and may be shared with the data repository. These samples could be used to research the causes of ISM, its complications and other conditions for which individuals with ISM are at increased risk, and to improve treatment. The repository will also be provided with a code-link that will allow linking the biological specimens with the phenotypic data from each participant, maintaining the blinding of the identity of the participant.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Participants With ISM: Patients who are currently being treated or plan to be treated for ISM

SUMMARY:
This is a Phase 4, non-interventional, observational study to collect detailed data on the clinical characteristics, clinical outcomes and medical management of ISM in real-world settings. The study will describe the demographic and clinical characteristics of ISM participants, including anaphylaxis and bone manifestations in ISM. Quality of life and disease control will be assessed through participant questionnaires. The study will also evaluate real world ISM treatment management, including use of avapritinib.

ELIGIBILITY:
Inclusion Criteria:

* Male or female adult participants (≥ 18 years of age) with a diagnosis of ISM according to the World Health Organization (WHO) diagnostic criteria
* Participant is currently being treated or plans to be treated with symptom-directed therapies and/or avapritinib for ISM.

Exclusion Criteria:

* Participants with advanced systemic mastocytosis (AdvSM) or another associated hematologic neoplasm
* Participants with smoldering systemic mastocytosis
* Ongoing participation in interventional studies in systemic mastocytosis (SM) at the time of enrollment
* Participants currently receiving treatment with a KIT inhibitor other than avapritinib at the time of enrollment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Participants with ISM who are currently being treated or plan to be treated with symptom-directed therapies and/or avapritinib for ISM.
Sampling Method: Non-Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2026-02-01 (Estimated); Primary Completion 2032-12-01 (Estimated); Study Completion 2032-12-01 (Estimated)

PRIMARY OUTCOMES:
Baseline Demographics | Baseline (Month 1)
Change From Baseline in Patient-Reported Outcomes Scores | Baseline up to Month 61
Change From Baseline in Serum KIT D816V Variant Allele Frequency (VAF) | Baseline up to Month 61
Change From Baseline in Serum Tryptase | Baseline up to Month 61
Change From Baseline in Indolent Systemic Mastocytosis (ISM) Symptom-Directed Therapies | Baseline up to Month 61